CLINICAL TRIAL: NCT06432972
Title: Accelerated Pulmonary Rehabilitation in the Preoperative Period
Acronym: PREHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Katherine Menson, Principal Investigator, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002705; 1143233 (Other Grant/Funding Number: American Lung Association)
Record Dates: First submitted 2024-05-13; First posted 2024-05-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Cancer
Keywords: Pulmonary Rehab
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehab (Experimental)
  Interventions: Other: Pulmonary Rehab

INTERVENTIONS:
Other: Pulmonary Rehab — Prehab will include 2, one-hour sequential sessions of PR per day as is standard, however this intervention will increase the frequency from 2 days to 4 days per week, for 2 weeks, thus completing 16 sessions of PR prior to surgery. An exercise prescription will be written by the medical director based on initial 6MWD, age, height, weight, and co-morbidities, as is standard of care. Prior to each session, patients are evaluated for symptoms and vital signs are measured. Exercise will include 30 minutes of warm-up and upper and lower extremity resistance training, either against gravity or with resistance bands as appropriate. Exercise will then move to the open gym, where patients utilize endurance equipment of their choosing, such as a treadmill or recumbent bicycle. As with traditional PR, participants will be given online education videos regarding lung health to complete at home, with a supplementary video on breathing techniques to reduce atelectasis from pain.

SUMMARY:
This proposed project will be a single arm, non-masked study. Participants who are actively smoking with a diagnosis of a new lung nodule, either confirmed or suspicious for lung cancer, with a plan for lung cancer treatment with or without surgical resection will be recruited from the University of Vermont Medical Center (UVMMC)pulmonary, cardiothoracic surgery, and Lung Multidisciplinary Clinic (LMDC). All patients will be enrolled in prehab and offered smoking cessation therapy. The acceptability and feasibility of this intervention will be measured by percent enrollment in study, attendance, barriers to completion, and monitoring of adverse events. The effect of prehab will be measured by traditional metrics, including fitness, respiratory symptoms, and depression scale. Research outcomes will be measured by smoking habits, anxiety, and surgical complications.

Investigators estimate that 20 participants over a two-year period will be sufficient to measure the safety and feasibility of this study. Investigators aim to enroll, on average, 2 participants per month in order to complete this study in a timely fashion. Participants will be enrolled in prehab on a rolling basis, as to not delay surgical timeline.

DETAILED DESCRIPTION:
The benefits of pulmonary rehab (PR) prior to lung resection have not been well-studied in the population that could benefit from it the most, patients with COPD who smoke. This study would be innovative in two major ways. First, the impact of prehab in those who smoke could be established. Secondly, the optimal model of prehab, which meets the clinical needs of the patient in the pre-surgical window, and aligns with the current model of PR, could be determined.

Screening and Recruitment Investigators estimate that 20 participants over a two-year period will be sufficient to measure the safety and feasibility of this study. Investigators aim to enroll, on average, 2 participants per month in order to complete this study in a timely fashion. Participants will be enrolled in prehab on a rolling basis, as to not delay surgical timeline.

Some procedures will be performed as a component of standard of care and some will be for research purposes only. This distinction is outlined in the sections below.

Intake and Baseline Assessment After informed consent, participants will complete the initial assessment with study coordinator. This will include anthropometrics, demographics like age, sex, race and ethnicity, and other sociodemographic and economic characteristics such as education, marital status, income, etc. This assessment will also include thorough medical, and surgical review, healthcare resource utilization, medication usage, substance use and smoking history, specifically recall of average cigarettes per day, carbon monoxide measurements, Fagerström nicotine dependence scale, and readiness to change. Investigators will also administer the General Anxiety Disorder-7 (GAD-7) questionnaire to assess for anxiety. Following intake, participants will be enrolled in the prehab program, which will include standard of care intake measurements including 6-minute walk distance (6MWD), mMRC, SGRQ, short physical performance battery (SPPB), and PHQ-9. For ease of the patient, Investigators will offer that this be performed on the same day, in a private medical setting at the PR facility. If the patient chooses, Investigators can offer intake at the Vermont Lung Center on a separate day.

Prehab Prehab will include 2, one-hour sequential sessions of PR per day as is standard, however this intervention will increase the frequency from 2 days to 4 days per week, for 2 weeks, thus completing 16 sessions of PR prior to or in the early stages of treatment. An exercise prescription will be written by the medical director based on initial 6MWD, age, height, weight, and co-morbidities, as is standard of care. Prior to each session, patients are evaluated for symptoms and vital signs are measured. Exercise will include 30 minutes of warm-up and upper and lower extremity resistance training, either against gravity or with resistance bands as appropriate. Exercise will then move to the open gym, where patients utilize endurance equipment of their choosing, such as a treadmill or recumbent bicycle. As with traditional PR, participants will be given online education videos regarding lung health to complete at home, with a supplementary video on breathing techniques to reduce atelectasis from pain. Virtual synchronous home-based PR will be offered to patients who have barriers to in-center PR.

Smoking Cessation Intervention Regarding smoking cessation, patients will be offered and prescribed the gold standard therapies in an attempt at smoking cessation, including a one-hour individual counseling session with a mental health therapist trained in smoking cessation therapy, varenicline treatment, dual acting NRT, and referral to the state smoking cessation program. Education modules on the benefits of smoking cessation will also be created for participants to review in the education portion of prehab. None of these interventions will be required, but offered as is standard of care.

Assessments Post-Prehab and 30 Days Post-Treatment Following completion of prehab prior to lung resection surgery Pulmonary Rehabilitation standard of care assessments and research-based assessments will be repeated. This will include interim health history, healthcare resource utilization, and medication usage, assessment for adverse events and COPD exacerbations, substance use and smoking status including recall of average cigarettes per day, carbon monoxide measurements, Fagerström nicotine dependence scale, readiness to change, GAD-7 and the study evaluation. 30 days following lung cancer treatment, the study team will review the participants medical record for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Lung nodule that is deemed highly suspicious for lung cancer based on: nodule characteristics, risk factors, CT-PET avidity, previous biopsy results, and assessment by physicians specializing in lung cancers
* Eligible for treatment
* Current cigarette smoking ≥5 cigarettes per day
* Willing to attempt smoking cessation during prehab period
* Willing to take nicotine replacement therapy (NRT) and varenicline
* Able to attend PR at UVMMC for 2, one-hour sequential sessions for a total of 16 sessions over 8 days in a 2-week time frame
* Willing and able to provide informed consent; ability determined by study physician and/or LMDC treatment physicians

Exclusion Criteria:

* Unable to safely participate in PR due to unstable cardiac disease, unstable peripheral vascular disease, musculoskeletal disease that would prevent exercise, significant psychiatric or neurocognitive disease that would limit ability to exercise safely in a group setting as determined by the study physician and/or treatment physicians
* Inability to consistently attend PR over a 2-week period
* Pregnancy, per patient self-report
* Active or recent participation in another clinical trial that, in the opinion of the investigator would impact outcomes measured in this study
* Any other condition in the opinion of the investigator/study physician and or treatment physicians that would jeopardize patient safety or integrity of research results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients determined eligible who enroll in the study | Through study completion, approximately 2 years
  Acceptability and feasibility will be documented by percent of those eligible enrolling in the study.
Average Pulmonary Rehab sessions completed | The 14 day (up to 21 day) intervention period
  Acceptability and feasibility will be determined by the proportion of pulmonary rehab sessions completed during this condensed pulmonary rehab program

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT06432972/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT06432972/ICF_001.pdf